CLINICAL TRIAL: NCT04100967
Title: Examination of Habitual Sleep Trajectories Across the First Two Years of College: Relation to Weight Gain Risk Behaviors and Outcomes
Brief Title: Examining the Longitudinal Relationship Between Sleep and Weight Gain in College Students
Acronym: STARLIT
Status: Completed | Type: Observational
Sponsor: Oakland University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 898494; 1R15HL130955-01A1 (NIH)
Record Dates: First submitted 2019-09-18; First posted 2019-09-24 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Healthy; Overweight
Keywords: sleep; obesity; body fat composition; young adults; diet; activity; Dual X-ray Absorptiometry
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This two-year prospective, observational study examines the relationship between habitual short sleep and weight gain, as well as the association between habitual short sleep and behaviors that put people at risk of weight gain. Habitual short sleep is defined as sleeping <6 hours per night on average. Participants will be healthy freshmen college students who are normal weight or overweight. Exclusion criteria include pregnancy, an inability to be ambulatory, currently taking a medication that could influence or interfere with sleep, or reporting a past/current neurological problem, past/current head injury, past/current sleep disorder, current mood, anxiety, or substance use disorder, current psychosis, or current suicidal ideation/plans. Recruitment will be during new student orientations that occur prior to fall semester. Eligibility will be determined using a screening interview, the DSM-5 Self-Rated Level 1 Cross-Cutting Symptom Measure - Adult, and DSM-5 Self-Rated Level 2 measures. Eligible participants will be assessed at baseline (time 1), and 8, 16, and 24 months after Time 1. Sleep, physical activity, food/beverages, substance use, and technology use will be collected daily during each eight day recording period. Sleep will be measured with a sleep monitor, activity will be assessed using an accelerometer, food/beverages will be obtained using the National Cancer Institute's Automated Self-Administered 24-hour Dietary Assessment Tool, and substance use and technology use will be measured via self-report. Participants will attend a session after each recording period to have weight and height measured, be scanned via Dual-energy x-ray absorptiometry (DXA), and complete a packet of questionnaires about demographics, health, sleep quality and beliefs, life events, food cravings, and physical development. It is hypothesized that participants will have different habitual sleep trajectories over time. It is also hypothesized that two particular sleep trajectories (stable habitual short sleep and increasingly shorter habitual sleep across time) will be significantly related to weight gain, increased body fat percent, and weight gain risk behaviors (i.e., increased caloric intake and decreased physical activity). Finally, it is hypothesized that the two sleep trajectories will be significantly associated with higher rates of media and technology use and higher rates of problematic sleep-related beliefs/behaviors.

ELIGIBILITY:
Inclusion Criteria:

* College freshmen
* Traditional college age
* BMI from 18.5-29.9.

Exclusion Criteria:

* Neurological problem
* Head injury
* Sleep disorder
* Mood disorder
* Anxiety disorder
* Substance use disorder
* Psychosis
* Suicidal ideation/plan
* Lacking the ability to be ambulatory
* Pregnancy

Ages: 17 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: College freshmen
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline total body fat percentage at 24 months | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea T. Kozak, PhD, Principal Investigator — Oakland University
Locations (1):
- Oakland University, Rochester, Michigan, United States

REFERENCES:
- [Derived] Kozak AT, Pickett SM, Jarrett NL, Markarian SA, Lahar KI, Goldstick JE. Project STARLIT: protocol of a longitudinal study of habitual sleep trajectories, weight gain, and obesity risk behaviors in college students. BMC Public Health. 2019 Dec 23;19(1):1720. doi: 10.1186/s12889-019-7697-x. PMID 31870336